CLINICAL TRIAL: NCT00703885
Title: PharmacofMRI of Anxiolytic Medications (Alprazolam)
Brief Title: PharmacofMRI (Functional Magnetic Resonance Imaging) of Anxiolytic Medications (Alprazolam)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Murray B. Stein, Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: UCSD IRB 060407 - A; R01MH075792 (NIH)
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Anxiety Disorders
Keywords: functional magnetic resonance imaging; fMRI; alprazolam; anxiety disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Alprazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 0.25 mg alprazolam PO (liquid) will be administered 1 hour prior to fMRI scan.
  One-time, single dose.
  Note that subjects receive all 3 treatments in randomized order (cross-over study), approximately 7-10 days apart.
  Interventions: Drug: 0.25 mg alprazolam
- 2 (Active Comparator): 1 mg alprazolam PO (liquid) will be administered 1 hour prior to fMRI scan
  One-time, single dose.
  Note that subjects receive all 3 treatments in randomized order (cross-over study), approximately 7-10 days apart.
  Interventions: Drug: 1.0 mg alprazolam
- Placebo (Placebo Comparator): Inactive ingredient in liquid matching appearance and volume of the two active alprazolam dose comparators.
  Note that subjects receive all 3 treatments in randomized order (cross-over study), approximately 7-10 days apart.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 0.25 mg alprazolam — 0.25 mg alprazolam PO (liquid) to be administered 1 hour prior to fMRI scan
  Note that subjects receive all 3 treatments in randomized order (cross-over study), approximately 7-10 days apart.
  Other Names: Xanax
  Arms: 1
Drug: 1.0 mg alprazolam — 1 mg alprazolam PO (liquid) will be administered 1 hour prior to fMRI scan
  Note that subjects receive all 3 treatments in randomized order (cross-over study), approximately 7-10 days apart.
  Other Names: Xanax
  Arms: 2
Drug: placebo — Placebo (liquid) to be administered 1 hour prior to fMRI scan
  Note that subjects receive all 3 treatments in randomized order (cross-over study), approximately 7-10 days apart.
  Arms: Placebo

SUMMARY:
The purpose of this study is to use functional magnetic resonance imaging (fMRI) in healthy controls to examine the acute effects of certain anxiolytic medications on brain function.

DETAILED DESCRIPTION:
Increased amygdala and insula activity have been implicated in neurobiological models of anxiety. Using fMRI, the anxiolytic medication, lorazepam, has previously been found to decrease activation in these areas during the processing of emotional stimuli. This study aims to replicate those results but by using a different medication, alprazolam. An eventual aim of this study, in combination with future studies, is to evaluate the utility of fMRI as a tool to identify anxiolytic function in both established and novel compounds that may be used to treat anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Male, or female (not pregnant or intending to become pregnant during the study)
* Between the ages of 18-30.
* In good general health.
* No specific contraindications to the drug being administered

Exclusion Criteria:

* Subjects with a history of DSM-IV depressive disorder, psychotic disorder, anxiety disorder
* Subjects who meet criteria for substance abuse or dependence within the last 6 months
* Subjects with an positive urine screen for illicit drugs
* having clinically significant abnormal laboratory, ECG or physical examination findings not resolved by the baseline visit
* Patients who have taken psychotropic drugs or antidepressants (including monoamine oxidase inhibitors, MAOI's) within the last year
* subject is left-handed.
* The subject suffers from claustrophobia, or phobia for injections or blood.
* Magnetic Resonance Imaging related exclusion criteria: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), subjects who have ever been a metal worker/welder; history of eye surgery/eyes washed out because of metal, aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, subjects who are in the first trimester of pregnancy, subjects with an I.U.D. (birth control device), a shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray B Stein, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Simmons AN, Arce E, Lovero KL, Stein MB, Paulus MP. Subchronic SSRI administration reduces insula response during affective anticipation in healthy volunteers. Int J Neuropsychopharmacol. 2009 Sep;12(8):1009-20. doi: 10.1017/S1461145709990149. Epub 2009 Jun 23. PMID 19545475
- [Background] Aupperle RL, Ravindran L, Tankersley D, Flagan T, Stein NR, Simmons AN, Stein MB, Paulus MP. Pregabalin influences insula and amygdala activation during anticipation of emotional images. Neuropsychopharmacology. 2011 Jun;36(7):1466-77. doi: 10.1038/npp.2011.32. Epub 2011 Mar 23. PMID 21430645
- [Background] Aupperle RL, Tankersley D, Ravindran LN, Flagan T, Stein NR, Stein MB, Paulus MP. Pregabalin effects on neural response to emotional faces. Front Hum Neurosci. 2012 Mar 27;6:42. doi: 10.3389/fnhum.2012.00042. eCollection 2012. PMID 22470326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects receive both doses of active drug and placebo in randomized order.
Pre-assignment Details: All subjects receive both doses of active drug and placebo in randomized order.
Groups:
- ALL SUBJECTS RECEIVE ALL 3 TREATMENTS: Alprazolam Low Dose Alprazolam High Dose Placebo
  Sequence of administration not available for subjects
Period: Overall Study
Arm/Group | ALL SUBJECTS RECEIVE ALL 3 TREATMENTS
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- ALL SUBJECTS RECEIVE ALL 3 TREATMENTS: Alprazolam Low Dose Alprazolam High Dose Placebo
  Please note that this is a cross-over design with all subjects receiving all three treatments
Arm/Group | ALL SUBJECTS RECEIVE ALL 3 TREATMENTS
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Effect of Alprazolam Versus Placebo on BOLD fMRI During Emotion Processing
Description: Analysis not completed.
Time Frame: Same Day
Groups:
- BOLD fMRI: Cross-over design. Each subject receives, on alternate days and in randomized fashion, either low dose, high dose, or placebo
Arm/Group | BOLD fMRI
Number analyzed (Participants) | 0

2. Primary Outcome: Voxelwise Brain Imaging Data
Description: Analysis of data not completed.
Time Frame: Post-Rx Administration
Groups:
- Imaging Data for Repeated Measures: Crossover design. Each subject receives, in randomized order and on different days:
  Low dose alprazolam High dose alprazolam Placebo
Arm/Group | Imaging Data for Repeated Measures
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Acute effects within 2 hours of drug administration
Description: Acute, single-dose study
Groups:
- ALL SUBJECTS RECEIVE ALL 3 TREATMENTS: Alprazolam Low Dose Alprazolam High Dose Placebo
Arm/Group | ALL SUBJECTS RECEIVE ALL 3 TREATMENTS
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
This is a single dose cross-over study in 16 healthy subjects.

BOLD fMRI analyses for this study were not completed by the investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No